CLINICAL TRIAL: NCT04868162
Title: An Open-Label, Single Arm, Multi-Center Phase II Clinical Study to Evaluate the Efficacy and Safety of MRG003 in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of Head and Neck.
Brief Title: A Study to Evaluate the Efficacy and Safety of MRG003 in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of Head and Neck
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG003-004
Record Dates: First submitted 2021-04-29; First posted 2021-04-30 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Recurrent or Metastatic Squamous Cell Carcinoma of Head and Neck
Keywords: MRG003; Squamous Cell Carcinoma of Head and Neck; EGFR; HX008; PD-1
MeSH Terms: conditions — Recurrence; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Arm (Experimental): MRG003 monotherapy will be administered for patients enrolled into Part A of this study; MRG003 and HX008 combination will be administered for patients enrolled into Part B of this study.
  Interventions: Drug: MRG003; Drug: MRG003+HX008

INTERVENTIONS:
Drug: MRG003 — On the first day of every 3 weeks, MRG003 will be administered via intravenous infusion at 2.0 mg/kg or 2.3 mg/kg.
Drug: MRG003+HX008 — On the first day of every 3 weeks, MRG003 will be administered via intravenous infusion at 2.0 mg/kg or the recommended dose by SMC; and HX008 will be administered via intravenous infusion at 3.0 mg/kg

SUMMARY:
The objective of this study is to assess the safety, efficacy, pharmacokinetics, and immunogenicity of MRG003 and the combination of MRG003 and HX008 in patients with recurrent or metastatic squamous cell carcinoma of head and neck.

DETAILED DESCRIPTION:
The study consists of two stages. In Part A, approximately 60 patients will be enrolled to evaluate the safety and preliminarily efficacy of MRG003 at 2.0 and 2.3 mg/kg, to further explore the optimized dose. In Part B, 30 to 50 patients will be enrolled to evaluate the safety and preliminary efficacy of the combination of MRG003 and HX008.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the ICF and follow the requirements specified in the protocol.
* Expected survival time≥3 months.
* Patients with histologically confirmed unresectable recurrent or metastatic squamous cell carcinoma of head and neck.
* Failed prior platinum and/or anti-PD-1 treatment (Part A); failed or intolerant to at least one prior line of standard therapy (platinum-based regimen) (Part B)
* Patients must have at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
* ECOG performance score 0 or 1.
* Organ functions and coagulation function must meet the basic requirements.
* Serum or urine pregnancy test negative within 7 days before the first dose of investigational drug.
* Patients with childbearing potential must use effective contraception during the treatment and for 6 months after the last dose of treatment.

Exclusion Criteria:

* History of 4 or more systemic anti-tumor therapies for the recurrent or metastatic squamous cell carcinoma of head and neck.
* ≥Grade 2 peripheral neuropathy
* Prior anti-tumor therapy with MMAE/MMAF ADCs
* BMI≤17
* Expected surgery or any other form of systemic or local anti-tumor therapy.
* History of systemic chemotherapy within 3 weeks before the first administration of the investigational drug, targeted small molecule therapy within 2 weeks or 5 half-life periods before the first administration (whichever is shorter), antitumor biological therapy or immunotherapy within 4 weeks before the first administration, or major surgery.
* Known active CNS metastasis and/or cancerous meningitis.
* Residual toxicity reactions caused by previous anti-tumor treatment or abnormal values of laboratory tests higher than grade 1 (CTCAE v5.0). Prior Grade 3 to 4 immune-related AE (irAE) or ≥Grade 2 heart-related irAE.
* Uncontrolled or poorly controlled heart disease.
* History of pulmonary embolism or deep vein thrombosis within 3 months before the first administration of the investigational drug.
* Known history of malignancy.
* History of severe dermatosis.
* Uncontrolled or poorly controlled hypertension.
* Patients with a history of active bleeding, coagulopathy, or receiving coumarin anticoagulation therapy.
* Known allergic reaction to any ingredients or excipients of investigational drugs.
* Known active hepatitis B or C.
* Complicated with severe, uncontrolled infection or known human immunodeficiency virus (HIV) infection, or diagnosed as acquired immunodeficiency syndrome (AIDS); or uncontrolled autoimmune disease; or history of allogeneic tissue/organ transplantation, stem cell or bone marrow transplantation, or solid organ transplantation.
* Active bacterial, viral, fungal, rickettsia, or parasitic infections that require systemic anti-infective treatment.
* Vaccination of live virus vaccine within 30 days before the first administration of the study drug. Inactivated seasonal influenza vaccine or approved COVID-19 vaccine is allowed.
* History of previous or concurrent interstitial pneumonia, radiation pneumonitis, severe chronic obstructive pulmonary disease, severe pulmonary dysfunction, symptomatic bronchospasm, etc.
* Patients receiving immunology-based treatment for any reason.
* Uncontrolled pleural effusion, pericardial effusion or recurrent ascites.
* Potent CYP3A4 inhibitors or inducers are in use and cannot be discontinued.
* Women who are lactating or pregnant.
* Other conditions that in the clinical judgement of the investigator make the patient not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by Investigator per RECIST v1.1 | Baseline to study completion (up to 24 months)
  ORR is defined as the proportions of patients with a complete response (CR) and partial response (PR). ORR will be assessed according to RECIST v1.1.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Baseline to study completion (up to 24 months)
  DCR is defined as the proportion of subjects achieving CR, PR, and stable disease (SD) after treatment.
Duration of Response (DoR) | Baseline to study completion (up to 24 months)
  The time interval between the date of the earliest qualifying response and the date of disease progression or death for any cause, whichever occurs earlier.
Progression Free Survival (PFS) as assessed by investigator | Baseline to study completion (up to 24 months)
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Overall Survival (OS) | Baseline to study completion (up to 24 months)
  OS is defined as the duration from the start of treatment to death of any cause.
Adverse Events (AEs) | Baseline to 30 days after the last dose of study treatment
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.
Serious Adverse Events (SAEs) | Baseline to 45 days after the last dose of study treatment
  Adverse events that are fatal, life-threatening, or result in hospitalization or prolonged hospitalization, persistent or significant disability/incapacity/substantial disruption of the ability to lead a normal life, congenital anomaly/birth defect or major medical events or reactions
Tmax | Baseline to 30 days after the last dose of study treatment
  Time to reach the maximum blood concentration
Cmax | Baseline to 30 days after the last dose of study treatment
  Maximum observed blood concentration
AUClast | Baseline to 30 days after the last dose of study treatment
  Area under the blood concentration-time curve from time 0 to the time of last quantifiable concentration
Incidence of anti-drug antibody (ADA) | Baseline to 30 days after the last dose of study treatment
  The proportion of patients with positive ADA immunogenicity results.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, Doctor, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No